CLINICAL TRIAL: NCT00324766
Title: Safety and Efficacy of Levosimendan in Patients With Acute Myocardial Infarction Complicated by Symptomatic Left Ventricular Failure.
Brief Title: Levosimendan in Acute Heart Failure Following Acute Myocardial Infarction.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0105
Record Dates: First submitted 2006-05-10; First posted 2006-05-11 (Estimated); Last update posted 2012-06-26 (Estimated); Status verified 2012-06

CONDITIONS: Myocardial Infarction; Heart Failure; Cardiogenic Shock
MeSH Terms: conditions — Myocardial Infarction; Heart Failure; Shock, Cardiogenic | interventions — Simendan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): levosimendan
  Interventions: Drug: levosimendan
- 2 (Placebo Comparator): Placebo, 1 h infusion, 0.2 microgs/kg/min, 24 h infusion,0.1 microgs/kg/min
  Interventions: Drug: placebo,

INTERVENTIONS:
Drug: levosimendan — 1 h infusion, 0.2 microgs/kg/min, 24 h infusion,0.1 microgs/kg/min
  Other Names: Simdax
  Arms: 1
Drug: placebo, — 24 h, infusion
  Other Names: placebo
  Arms: 2

SUMMARY:
The purpose of this study is to determine the safety and efficacy of a 24 hour infusion with levosimendan in patients with acute myocardial infarction and heart failure after acute percutaneous coronary intervention (PCI) treatment.

DETAILED DESCRIPTION:
Double blind placebo-controlled study with parallel groups in patients with acute PCI treated myocardial infarction complicated with decompensated heart failure. The study include a prospectively defined subgroup of patients in cardiogenic shock. Treating acute myocardial infarction with PCI restores blood flow, but decreased contractility remains for hours and days due to stunned myocardium. Levosimendan has both inotropic and vasodilatory effects which could support the failing heart after treating the acute myocardial infarction with PCI and may improve myocardial stunning and decrease pro-inflammatory cytokines. Levosimendan could improve myocardial contractility, symptoms and outcome without adverse effects. The aims of the study are to investigate whether a 24 hour infusion with levosimendan could improve regional contractility measured by echocardiography, improve BNP levels, reduce the levels of pro-inflammatory cytokines and improve symptoms in patients with acute decompensated heart failure during the first 24 hours after acute PCI.

ELIGIBILITY:
Inclusion Criteria:

* Acute ST-elevation myocardial infarction subject to acute PCI or non-ST elevation myocardial infarction subject to PCI within 72 hours after start of chest pain and:
* Revascularization by PCI,
* Signs of decreased wall-motion in at least 3 of 16 segments of the left ventricle
* Dyspnoea at rest and one of the following:

pulmonary edema, pulmonary congestion,need for CPAP or ventilator, need for IC diuretics or oliguria.

Subgroup of patients in cardiogenic shock: Systolic BP below 90 after 1 hour of volume therapy.

Exclusion Criteria:

* Age below 20 years
* Heart rate above 120 bpm
* Septic shock
* ARDS
* Creatinine >450 micromol/l
* Hepatic impairment
* Significant mechanical outlet obstruction
* Allergy against study drug medication
* Anaemia (Hb <8 g/dl)
* Pregnancy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2006-06; Primary Completion 2011-09 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Efficacy: Changes in regional contractility measured as wall-motion score index, proBNP and clinical symptoms. | At 5 days
  Changes in regional contractility (WMSI) measured by echo is the primary endpoint in the study and the sample size calculation is based on expected differenced in WMSI from baseline to day 5 between groups.

SECONDARY OUTCOMES:
Mace: Time to death, non-fatal myocardial infarction or revascularization during the first 6 weeks and 6 months. | 6 months
Time to rehospitalisation for decompensated heart failure. | 6 months
Days hospitalised/days in intensive/coronary care. | At discharge
Changes in inflammation markers. | 1, 5 days, 6 weeks.
Improvement in creatinine clearance. | 5 days
Improvement of hemodynamic parameters. | 5 days
Central venous oxygen saturation. | 1 day
Total mortality. | 6 months
Arrhythmias, hypotension, ischaemic episodes. | 5 days
Change in proBNP | Baseline to day 5
Change in clinical symptom score | Baseline to day 5

CONTACTS AND LOCATIONS:
Overall Officials: Trygve Husebye, MD,, Principal Investigator — Department of Cardiology, Ulleval University Hospital; Geir Ø Andersen, MD, PhD, Study Chair — Department of Cardiology, Ulleval University Hospital
Locations (1):
- Department of Cardiology, Ulleval University Hospital, Oslo, Norway

REFERENCES:
- [Derived] Langseth MS, Andersen GO, Husebye T, Arnesen H, Zucknick M, Solheim S, Eritsland J, Seljeflot I, Opstad TB, Helseth R. Neutrophil extracellular trap components and myocardial recovery in post-ischemic acute heart failure. PLoS One. 2020 Oct 29;15(10):e0241333. doi: 10.1371/journal.pone.0241333. eCollection 2020. PMID 33119664
- [Derived] Husebye T, Eritsland J, Arnesen H, Bjornerheim R, Mangschau A, Seljeflot I, Andersen GO. Association of interleukin 8 and myocardial recovery in patients with ST-elevation myocardial infarction complicated by acute heart failure. PLoS One. 2014 Nov 12;9(11):e112359. doi: 10.1371/journal.pone.0112359. eCollection 2014. PMID 25390695
- [Derived] Husebye T, Eritsland J, Muller C, Sandvik L, Arnesen H, Seljeflot I, Mangschau A, Bjornerheim R, Andersen GO. Levosimendan in acute heart failure following primary percutaneous coronary intervention-treated acute ST-elevation myocardial infarction. Results from the LEAF trial: a randomized, placebo-controlled study. Eur J Heart Fail. 2013 May;15(5):565-72. doi: 10.1093/eurjhf/hfs215. Epub 2013 Jan 2. PMID 23288914